CLINICAL TRIAL: NCT05350644
Title: Predicting Response to Medical Treatment of Inflammatory Bowel Disease (IBD) Using Single Cell Transcriptomic on Intestinal Biopsies: a Prospective Cohort Study of Personalized Medicine
Brief Title: Inflammatory Bowel Disease(IBD), Treatment Response
Status: Terminated | Type: Observational
Why Stopped: Recruitment of patients for this clinical trial has been withdrawn due to logistical challenges and the inability to enroll a sufficient number of participants meeting the specific eligibility criteria within the projected timeline.
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Hospital of Southern Jutland (Other); University of Kiel (Other); Colitis-Crohn Foreningen (Other)
Responsible Party: Principal Investigator, Vibeke Andersen, Professor, University of Southern Denmark
Other Study IDs: BELIEVE-IBD-SCT
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2022-05

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
Keywords: Biomarkers; Treatment outcome; Transcriptomics
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Intestinal biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Primary exposure variable — 1. Specific activated CD8+ T-cell transcriptome signature in biopsies is associated with better treatment outcome
  2. Specific activated CD8+ T-cell transcriptome signature in blood is associated with better treatment outcome
  Other Names: Transcriptome signature
Other: Other (exploratory) exposure variables — Specific transcriptomic signatures in intestinal biopsies and peripheral blood mononuclear cells (PBMCs) of IBD patients can work as a predictive biomarker for the tumor necrosis factor inhibitors (TNFi) treatment response

SUMMARY:
Inflammatory bowel diseases (IBD) is treated with biologics targeting the pro-inflammatory molecule tumour necrosis factor-α (TNF), i.e. TNF inhibitors. Up to one third of the patients do, however, not respond to biologics and little is known of the biological mechanism as a prognostic factor (possibly enabling personalised medicine). The aim of this project is to identify biomarkers that support individualized forecasting of optimized treatment outcome on these costly drugs.

This prospective cohort study will enroll IBD patients assigned for biologic treatment. At baseline (Pre-treatment), biopsies and blood is taken from each patient. Follow-up will be conducted at week 14-16 after treatment initiation (according to the current Danish standards). Evaluation of a successful treatment outcome response will - for each disease - be based on most frequently used primary endpoints; the major outcome of the analyses will be to detect differences in treatment outcome between patients with the cell expression.

The overarching goal of this project is to improve the lives of patients suffering from IBD, by providing evidence to potential biomarkers that would be likely to improve the clinical outcome.

The study is approved by the local Ethics Committee (S-20160124) and the local Data Agency (2008-58-035). The study findings will be disseminated in peer-reviewed journals, via patient associations, and presented at national and international conferences.

DETAILED DESCRIPTION:
Inflammatory bowel diseases [IBD] (of which Crohn's disease (CD) and ulcerative colitis (UC) are the two most prevailed entities) is a disease of the immune system that are managed with biological agents targeting the pro-inflammatory cytokine tumour necrosis factor-α (TNF), i.e. TNF inhibitors.

Design: In this prospective cohort study disease activity prior to and after (14-16 weeks) initiation of biologic treatment will be assessed. The endpoint is the treatment outcome defined as A: Responder according to the specific criteria described below (incl. drug-continuation) or B: Non-responder (incl. drug-discontinuation due to unacceptable side effects). Whether a patient will discontinue therapy is assumed to be based on a certain degree of shared decision making between the patient and physician supported by principles from national guidelines for each patient as recommended in the respective national guidelines and laboratory data.

Setting: All patients assigned for initiation of biologic treatment at the Department of Medical Gastroenterology, Odense University Hospital from 1st of February 2022 and until 31th of December 2022 or until a minimum of 20 patients with IBD is achieved.

Clinical data consist of personal data, data on health and disease and disease activity scores. Information registered by clinicians and technicians will be transferred from paper format to electronic format using either double entry of data or automated forms processing.

Sample size considerations: We will include a limited set of patient biopsies from 20 UC patients and analyze the changes in responders versus non-responders for identifying potential predictive pathways and biomarkers. Such a strategy has recently been proven valuable for identification of biomarkers predictive of treatment response in CD with a similar number of samples as in our study All data analysis will be done in R, transparently reporting the source code used to analyze the data.

Project organization: The project is organized with a Clinical Research Group and an Analytical Research Group. The clinical group includes specialists from the medical, gastroenterological, departments that are sampling the cohort. The analytical group will perform the analyses on the biological material.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with inflammatory bowel disease
* initiation of targeted therapy
* able to read and understand Danish

Exclusion Criteria:

* Patients with cancer
* Not mentally able to reply the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: targeted therapy and able to read and understand Danish.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
1. Clinical response to therapy depending on condition | week 14-16
  The predefined primary endpoint will be the proportion of patients with clinical response to therapy at first clinical follow-up.
  * Crohn's disease: Harvey Bradshaw Index (HBI) 4 or less (clinical remission) to <16 (non-remission)
  * Ulcerative colitis: Mayo Clinic Score of 2 or less (with no individual subscore of >1) (remission) to <12 (non-remission)

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Andersen, Prof, Principal Investigator — University of Southern Denmark
Locations (1):
- Odense University Hospital, Odense, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No